CLINICAL TRIAL: NCT07178795
Title: A Randomized Controlled Phase III Clinical Study of BL-M07D1 vs Pembrolizumab-platinum Chemotherapy in First-line Treatment of HER2-mutant Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study of BL-M07D1 vs Pembrolizumab-platinum Chemotherapy in First-line Treatment of HER2-mutant Advanced or Metastatic Non-squamous NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-306
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1
- Pembrolizumab-platinum chemotherapy (Active Comparator): Participants receive Pembrolizumab+Pemetrexed+Carboplatin or Cisplatin in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: BL-M07D1
Drug: Pembrolizumab — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Pembrolizumab-platinum chemotherapy
Drug: Pemetrexed — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Pembrolizumab-platinum chemotherapy
Drug: Carboplatin — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Pembrolizumab-platinum chemotherapy
Drug: Cisplatin — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Pembrolizumab-platinum chemotherapy

SUMMARY:
This trial is a registrational phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-M07D1 in patients with first-line treatment of HER2-mutant advanced or metastatic non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. Age at the time of signing the informed consent form is ≥18 years and ≤75 years, regardless of gender;
3. Expected survival time ≥12 weeks;
4. Histologically or cytologically confirmed advanced or metastatic non-squamous non-small cell lung cancer;
5. HER2 functional mutation confirmed by a central laboratory;
6. Provide the most recent tumor tissue meeting the requirements for biomarker testing by the central laboratory;
7. Must have at least one measurable target lesion as defined by RECIST v1.1;
8. ECOG performance status score of 0 or 1;
9. Toxicity from previous anti-tumor treatments has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. Organ function levels must meet the requirements;
11. For premenopausal women with childbearing potential, a pregnancy test must be conducted within 7 days prior to the start of treatment, and the serum pregnancy test must be negative. They must not be breastfeeding. All enrolled patients (regardless of gender) should take adequate and highly effective contraceptive measures throughout the treatment period and for 7 months after the end of treatment.

Exclusion Criteria:

1. Having undergone surgical treatment, radical radiotherapy, immunotherapy, etc., within 4 weeks prior to the first dose or within 5 half-lives;
2. Pathological findings indicating non-small cell carcinoma containing small cell carcinoma components and sarcomatoid carcinoma;
3. Concurrent presence of other driver gene mutations for which targeted drug therapy is available and approved for NSCLC indications;
4. Previous treatment with HER2-targeted therapy or ADC drugs with camptothecin derivatives as the toxin;
5. History of severe cardiovascular or cerebrovascular diseases within the past 6 months prior to screening;
6. Concurrent pulmonary diseases leading to severe impairment of lung function;
7. History of ILD/interstitial pneumonia requiring steroid treatment or current diagnosis of ILD/interstitial pneumonia;
8. Prolonged QT interval, complete left bundle branch block, third-degree atrioventricular block, frequent and uncontrollable arrhythmias;
9. Diagnosis of other primary malignancies within 5 years prior to the first dose;
10. Newly developed deep vein thrombosis within 14 days prior to screening;
11. Hypertension poorly controlled by antihypertensive medications;
12. Patients with central nervous system (CNS) metastases, carcinomatous meningitis (leptomeningeal metastases), and/or spinal cord compression;
13. Patients with a history of severe allergies to any excipients or components of the investigational drug;
14. History of autologous or allogeneic stem cell transplantation or organ transplantation;
15. Positive human immunodeficiency virus antibody, active hepatitis B virus infection, liver cirrhosis, or hepatitis C virus infection;
16. Occurrence of severe infections within 4 weeks prior to the first use of the investigational drug;
17. Patients with significant serous cavity effusion, symptomatic serous cavity effusion, or poorly controlled serous cavity effusion;
18. Systemic corticosteroid treatment with >10 mg/d prednisone or equivalent prior to randomization;
19. Presence of severe neurological or psychiatric disorders;
20. Subjects with clinically significant bleeding or obvious bleeding tendencies within 4 weeks prior to signing informed consent;
21. Conditions such as intestinal obstruction, Crohn's disease, ulcerative colitis, or chronic diarrhea;
22. Subjects planning to receive or having received live vaccines within 28 days prior to the first dose;
23. Presence of other severe physical or laboratory abnormalities, poor compliance, or any other factors that may increase the risk of participation in the study, interfere with study results, or make the patient unsuitable for participation in the study as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China